CLINICAL TRIAL: NCT03674684
Title: Rotational Thromboelastometry (ROTEM) Assessment of Modern Crystalloid, Hydroxyethyl Starch and Gelatin Effect on Coagulation in Vivo
Brief Title: ROTEM Assessment of Modern Crystalloid, Hydroxyethyl Starch and Gelatin Effect on Coagulation
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Durila Miroslav MUDr. Ph.D., associated professor, University Hospital, Motol
Other Study IDs: 14092018 Motol Hospital
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Coagulopathy
Keywords: hydroxyethyl starch, gelatin, ROTEM, coagulation
MeSH Terms: conditions — Hemostatic Disorders; Thrombosis | interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- hydroxyethyl starch: Patients who received hydroxyethyl starch
  Interventions: Other: hydroxyethyl starch
- gelatin: Patients who received gelatin
  Interventions: Other: hydroxyethyl starch
- crystalloids: Patients who received crystalloids
  Interventions: Other: hydroxyethyl starch

INTERVENTIONS:
Other: hydroxyethyl starch — After induction to anaesthesia patients received either hydroxyethyl starch or gelatin or crystalloids

SUMMARY:
Modern crystalloid and colloid solutions are balanced solutions which are increasingly used in perioperative period. However, studies investigating their negative effect on whole blood coagulation are missing. The aim of our study was to assess the effect of modern balanced crystalloid and colloid solutions on whole blood coagulation in vivo using rotational thromboelastometry.

DETAILED DESCRIPTION:
Blood samples were obtained from 30 patients during knee arthroscopy before and after administration of 500 ml of modern balanced crystalloid, hydroxyethyl starch (HES) or gelatin. Rotational thromboelastometry (EXTEM, INTEM and FIBTEM tests) were performed to assess negative effect of fluid solutions on whole blood coagulation.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients undergoing knee arthroscopy

Exclusion Criteria:

* receiving antiplatelet drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy patients undergoing knee arthroscopy
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-07-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
thromboelastometry assessment of coagulation | 3 months
  ROTEM tests- clotting time in seconds, Maximal clot firmness in mm, alpha angle of in degree of following tests EXTEM, INTEM, FIBTEM

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Durila, Principal Investigator — Second Medical Faculty, Charles University and University Hospital Motol
Locations (1):
- University Hopital Motol, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sevcikova S, Durila M, Vymazal T. [Rotational thromboelastometry assessment of ballanced crystalloid, hydroxyethyl starch and gelatin effects on coagulation: a randomized trial]. Braz J Anesthesiol. 2019 Jul-Aug;69(4):383-389. doi: 10.1016/j.bjan.2019.03.009. Epub 2019 Aug 9. PMID 31405567